CLINICAL TRIAL: NCT01044862
Title: Assessment of Multiple Intrauterine Gestations From Ovarian Stimulation
Acronym: AMIGOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pennsylvania (Other); University of Texas (Other); University of Vermont (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Heping Zhang, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMN-AMIGOS; 3U10HD055925-02S1 (NIH); 5U10HD055925 (NIH); 3U10HD039005-08S1 (NIH); 5U10HD039005 (NIH)
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Pregnancy; Unexplained Infertility
Keywords: Pregnancy; Infertility; Ovarian stimulation; Aromatase inhibitors; Follicle Stimulating Hormone
MeSH Terms: conditions — Infertility | interventions — Letrozole; Aromatase Inhibitors; Clomiphene; Follicle Stimulating Hormone; Gonadotropins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aromatase Inhibitors (AI) (Active Comparator): A daily dose of 5 mg of the AI, letrozole, will be administered orally for five days starting on day three of the menstrual cycle. Future cycles can be started at 2.5-7.5 mg/d. FDA approval (IND) will be obtained.
  Interventions: Drug: Letrozole (aromatase inhibitor)
- Clomiphene Citrate (CC) (Active Comparator): CC will be administered at a dose of 100 mg/d on cycle days 3-7. Future cycles can be started at 50-150 mg/d.
  Interventions: Drug: Clomiphene Citrate
- Follicle Stimulating Hormone (FSH) (Active Comparator): A daily injection of 150 IU of FSH will be administered subcutaneously starting on day three of the menstrual cycle and continuing until the day of hCG administration. Dosage will be able to be increased or decreased 37.5-75 IU/d beginning cycle day 7. Future cycles can be started at doses ranging from 75-225 IU/d. The same type of FSH injections will be used.
  Interventions: Drug: Follicle Stimulating Hormone (gonadotropin)

INTERVENTIONS:
Drug: Letrozole (aromatase inhibitor) — A daily dose of 5 mg of the AI, letrozole, will be administered orally for five days starting on day three of the menstrual cycle. Future cycles can be started at 2.5-7.5 mg/d. FDA approval (IND) will be obtained.
  Arms: Aromatase Inhibitors (AI)
Drug: Clomiphene Citrate — CC will be administered at a dose of 100 mg/d on cycle days 3-7. Future cycles can be started at 50-150 mg/d.
  Arms: Clomiphene Citrate (CC)
Drug: Follicle Stimulating Hormone (gonadotropin) — A daily injection of 150 IU of FSH will be administered subcutaneously starting on day three of the menstrual cycle and continuing until the day of hCG administration. Dosage will be able to be increased or decreased 37.5-75 IU/d beginning cycle day 7. Future cycles can be started at doses ranging from 75-225 IU/d. The same type of FSH injections will be used.
  Arms: Follicle Stimulating Hormone (FSH)

SUMMARY:
The objective of this application is to identify a pharmacologic agent which helps couples in whom the female partner ovulates regularly successfully obtain their goal of delivering a healthy child, whose use will result in low rates of multiple gestations. The central hypothesis is that, in infertile ovulatory women undergoing ovarian stimulation (OS) and intrauterine insemination (IUI), the use of aromatase inhibitors (AI) will stimulate the ovaries sufficiently to produce no reduction in the rate of pregnancy, while significantly reducing the numbers of multiple gestational pregnancies that result from stimulation with clomiphene citrate (CC) or follicle stimulating hormone (FSH). The rationale for the proposed research is that reduction of multiple pregnancy rates could significantly reduce maternal and neonatal morbidity and mortality, as well as the cost of healthcare for these individuals and society.

DETAILED DESCRIPTION:
Patient Population

The population will consist of 900 women up to and including women ≥18 to ≤40 years years of age (at time of randomization) desirous of conceiving who will be recruited over approximately a two year period from the Reproductive Medicine Network (RMN) clinical sites and possibly from the Specialized Cooperative Center Programs in Reproductive Research (SCCPIR) sites, through public notification programs.

Study Design

This will be a multi-center, prospective, partially blinded clinical trial of gonadotropins vs. clomiphene citrate vs. aromatase inhibitors. The randomization scheme will be coordinated through the data coordination center (DCC) and the randomization will be stratified by each participating site and within each site for ages 18-34 and 35-40.

Treatment

Patients will be randomized to receive either FSH, CC, or an AI according to randomization tables generated by a computer randomization program. Treatment assignments will be blocked by site and age group. Subjects randomized to pill treatment will receive medication in double blinded fashion, receiving one type of pill (overcoated CC or AI). Subjects randomized to injectable medication(FSH) will receive vials of medication.

Primary efficacy parameter

Multiple gestation rate following recruitment of multiple follicular development with an AI, as compared to CC and FSH.

Secondary efficacy parameters

Rate of pregnancy obtained, live birth rate, and time to pregnancy following administration of an aromatase inhibitor, as compared to CC and FSH as well as the live birth rate of multiple gestation pregnancies.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 to ≤40 years of age, with one or more years infertility history, desirous of conceiving, regularly ovulating (defined as 9 or more menses per year), at initiation of participation.
2. Normal uterine cavity and at least one open fallopian tube confirmed by hysterosalpingography (HSG), sonohysterography, or laparoscopy/hysteroscopy in the last three years preceding enrollment into the study. An uncomplicated intrauterine non-IVF pregnancy and uncomplicated delivery and postpartum course resulting in live birth within the last three years will also serve as sufficient evidence of a patent tube and normal uterine cavity as long as the subject did not have, during the pregnancy or subsequently, risk factors for Asherman's syndrome or tubal disease or other disorder leading to an increased suspicion for intrauterine abnormality or tubal occlusion.
3. Evidence of ovarian function/reserve as assessed by day 3 (+/-2 days) FSH ≤12 IU/L within one year prior to study initiation.
4. Normal or corrected thyroid function within one year of study initiation.
5. Normal prolactin level within one year of study initiation.
6. In general good health, not taking any medications which could interfere with the study (e.g., FSH, insulin sensitizers).
7. Ability to have inseminations following hCG administration.
8. Male partner with total motile sperm in the ejaculate of at least 5 million sperm, within one year of study initiation.

Exclusion Criteria:

1. Currently pregnant or successful pregnancies within 12 months of initiating participation. Clinical intrauterine miscarriages prior to initiating participation, within ASRM guidelines: subjects over 35 must wait six months, while subjects under 35 must wait 12 months. No exclusion for biochemical pregnancies.
2. Undiagnosed abnormal uterine bleeding.
3. Suspicious ovarian mass.
4. Patients on oral contraceptives, depo-progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive forms or implants, especially when the implants are still in place. A one-month washout will be required for patients on oral cyclic progestins.
5. Known 21-hydroxylase deficiency or other enzyme defect causing congenital adrenal hyperplasia.
6. Type I or Type II diabetes mellitus, or if receiving antidiabetic medications.
7. Known significant anemia (Hemoglobin <10 g/dL).
8. History of deep venous thrombosis, pulmonary embolus, or cerebrovascular event.
9. Known heart disease (New York Heart Association Class II or higher).
10. Known Liver disease (defined as AST or ALT>2 times normal, or total bilirubin >2.5 mg/dL).
11. Known Renal disease (defined as BUN >30 mg/dL or serum creatinine > 1.4 mg/dL).
12. History of, or suspected cervical carcinoma, endometrial carcinoma or breast carcinoma.
13. History of alcohol abuse (defined as >14 drinks/week) or binge drinking of ≥ 6 drinks at one time).
14. Known Cushing's disease.
15. Known or suspected adrenal or ovarian androgen secreting tumors.
16. Allergy or contraindication to the treatment medications: AI, gonadotropins, CC or hCG.
17. Couples with previous sterilization procedures (e.g. vasectomy, tubal ligation) which have been reversed.
18. Patients with untreated poorly controlled hypertension defined as a systolic blood pressure ≥ 160 mm Hg or a diastolic ≥ 100 mm Hg obtained on two measures obtained at least 60 minutes apart.
19. Subjects who have undergone a bariatric surgery procedure in the recent past (< 12 months) and are in a period of acute weight loss or have been advised against pregnancy by their bariatric surgeon.
20. Known moderate or severe endometriosis
21. Known polycystic ovarian syndrome as evidenced by anovulation or oligoovulation, hirsutism and/or elevated testosterone levels, and ovarian morphology on ultrasound examination.
22. Donated semen.
23. Couples in which either partner is legally married to someone else.
24. Medical conditions that are contraindications to pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2010-06; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — Albert Einstein College of Medicine; Michael Diamond, MD, Principal Investigator — Wayne State University; Richard Legro, MD, Study Director — Pennsylvania State University College of Medicine; William Schlaff, MD, Study Director — University of Colorado Denver Health Science Center; Gregory Christman, MD, Study Director — University of Michigan; Christos Coutifaris, MD, Study Director — University of Pennsylvania; Robert Brzyski, MD, PhD, Study Director — The University of Texas Health Science Center at San Antonio; Peter Casson, MD, Study Director — University of Vermont; Heping Zhang, PhD, Study Director — Yale University
Locations (14):
- United States (14):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Kuokkanen S, Seungdamrong A, Santoro N, Lieman H, Sun F, Wild R, Zhang H, Pal L. A relook at the relevance of thyroid stimulating hormone and thyroid autoimmunity for pregnancy outcomes: Analyses of randomized control trials data from Pregnancy in Polycystic Ovary Syndrome and Assessment of Multiple Intrauterine Gestations from Ovarian Stimulation. Fertil Steril. 2025 May;123(5):873-882. doi: 10.1016/j.fertnstert.2024.12.005. Epub 2024 Dec 12. PMID 39672366
- [Derived] Hosseinzadeh P, Peck JD, Burks HR, Souter I, Xing A, Craig LB, Diamond MP, Hansen KR. Follicular phase length is not related to live birth outcome in women with unexplained infertility undergoing ovarian stimulation with intrauterine insemination cycles in a multicenter trial. F S Rep. 2023 Aug 8;4(4):361-366. doi: 10.1016/j.xfre.2023.08.003. eCollection 2023 Dec. PMID 38204957
- [Derived] Gavrizi SZ, Arya S, Peck JD, Knudtson JF, Diamond MP, Wild RA, Hansen KR. High-sensitivity C-reactive protein levels and pregnancy outcomes in women with unexplained infertility after ovarian stimulation with intrauterine insemination in a multicenter trial. F S Rep. 2022 Jan 11;3(1):57-62. doi: 10.1016/j.xfre.2022.01.001. eCollection 2022 Mar. PMID 35386508
- [Derived] Souter I, Sun F, Zhang H, Diamond MP, Legro RS, Wild RA, Hansen KR, Santoro N; Eunice Kennedy Schriver National Institute of Child Health and Human Development Reproductive Medicine Network. A personalized medicine approach to ovulation induction/ovarian stimulation: development of a predictive model and online calculator from level-I evidence. Fertil Steril. 2022 Feb;117(2):408-418. doi: 10.1016/j.fertnstert.2021.10.024. PMID 35125179
- [Derived] Eisenberg E, Legro RS, Diamond MP, Huang H, O'Brien LM, Smith YR, Coutifaris C, Hansen KR, Santoro N, Zhang H. Sleep Habits of Women With Infertility. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4414-e4426. doi: 10.1210/clinem/dgab474. PMID 34180998
- [Derived] Engmann L, Sun F, Legro RS, Diamond MP, Zhang H, Santoro N; Reproductive Medicine Network. Factors associated with study protocol adherence and bio banking participation in reproductive medicine clinical trials and their relationship to live birth. Hum Reprod. 2020 Dec 1;35(12):2819-2831. doi: 10.1093/humrep/deaa232. PMID 33190149
- [Derived] Quaas AM, Gavrizi SZ, Peck JD, Diamond MP, Legro RS, Robinson RD, Casson P, Christman GM, Zhang H, Hansen KR; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Endometrial thickness after ovarian stimulation with gonadotropin, clomiphene, or letrozole for unexplained infertility, and association with treatment outcomes. Fertil Steril. 2021 Jan;115(1):213-220. doi: 10.1016/j.fertnstert.2020.07.030. Epub 2020 Sep 21. PMID 32972733
- [Derived] Kaing A, Jaswa EA, Diamond MP, Legro RS, Cedars MI, Huddleston HG. Highly elevated level of antimullerian hormone associated with preterm delivery in polycystic ovary syndrome patients who underwent ovulation induction. Fertil Steril. 2021 Feb;115(2):438-446. doi: 10.1016/j.fertnstert.2020.06.015. Epub 2020 Sep 1. PMID 32883514
- [Derived] Wang ET, Diamond MP, Alvero R, Casson P, Christman GM, Coutifaris C, Hansen KR, Sun F, Legro RS, Robinson RD, Usadi RS, Pisarska MD, Santoro NF, Zhang H; National Institute of Child Health and Human Development (NICHD) Reproductive Medicine Network. Androgenicity and fertility treatment in women with unexplained infertility. Fertil Steril. 2020 Mar;113(3):636-641. doi: 10.1016/j.fertnstert.2019.10.034. PMID 32192596
- [Derived] Trussell JC, Coward RM, Santoro N, Stetter C, Kunselman A, Diamond MP, Hansen KR, Krawetz SA, Legro RS, Heisenleder D, Smith J, Steiner A, Wild R, Casson P, Coutifaris C, Alvero RR, Robinson RB, Christman G, Patrizio P, Zhang H, Lindgren MC; Reproductive Medicine Network. Association between testosterone, semen parameters, and live birth in men with unexplained infertility in an intrauterine insemination population. Fertil Steril. 2019 Jun;111(6):1129-1134. doi: 10.1016/j.fertnstert.2019.01.034. Epub 2019 Apr 12. PMID 30982604
- [Derived] Barrett ES, Vitek W, Mbowe O, Thurston SW, Legro RS, Alvero R, Baker V, Bates GW, Casson P, Coutifaris C, Eisenberg E, Hansen K, Krawetz S, Robinson R, Rosen M, Usadi R, Zhang H, Santoro N, Diamond M. Allostatic load, a measure of chronic physiological stress, is associated with pregnancy outcomes, but not fertility, among women with unexplained infertility. Hum Reprod. 2018 Sep 1;33(9):1757-1766. doi: 10.1093/humrep/dey261. PMID 30085177
- [Derived] Butts SF, Seifer DB, Koelper N, Senapati S, Sammel MD, Hoofnagle AN, Kelly A, Krawetz SA, Santoro N, Zhang H, Diamond MP, Legro RS; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Vitamin D Deficiency Is Associated With Poor Ovarian Stimulation Outcome in PCOS but Not Unexplained Infertility. J Clin Endocrinol Metab. 2019 Feb 1;104(2):369-378. doi: 10.1210/jc.2018-00750. PMID 30085176
- [Derived] Evans-Hoeker EA, Eisenberg E, Diamond MP, Legro RS, Alvero R, Coutifaris C, Casson PR, Christman GM, Hansen KR, Zhang H, Santoro N, Steiner AZ; Reproductive Medicine Network. Major depression, antidepressant use, and male and female fertility. Fertil Steril. 2018 May;109(5):879-887. doi: 10.1016/j.fertnstert.2018.01.029. PMID 29778387
- [Derived] Hansen KR, Eisenberg E, Baker V, Hill MJ, Chen S, Talken S, Diamond MP, Legro RS, Coutifaris C, Alvero R, Robinson RD, Casson P, Christman GM, Santoro N, Zhang H, Wild RA; NICHD Reproductive Medicine Network. Midluteal Progesterone: A Marker of Treatment Outcomes in Couples With Unexplained Infertility. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2743-2751. doi: 10.1210/jc.2018-00642. PMID 29767754
- [Derived] Seungdamrong A, Steiner AZ, Gracia CR, Legro RS, Diamond MP, Coutifaris C, Schlaff WD, Casson P, Christman GM, Robinson RD, Huang H, Alvero R, Hansen KR, Jin S, Eisenberg E, Zhang H, Santoro N; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Preconceptional antithyroid peroxidase antibodies, but not thyroid-stimulating hormone, are associated with decreased live birth rates in infertile women. Fertil Steril. 2017 Oct 25:S0015-0282(17)31748-X. doi: 10.1016/j.fertnstert.2017.08.026. Online ahead of print. PMID 29102040
- [Derived] Styer AK, Jin S, Liu D, Wang B, Polotsky AJ, Christianson MS, Vitek W, Engmann L, Hansen K, Wild R, Legro RS, Coutifaris C, Alvero R, Robinson RD, Casson P, Christman GM, Christy A, Diamond MP, Eisenberg E, Zhang H, Santoro N; National Institute of Child Health and Human Development Reproductive Medicine Network. Association of uterine fibroids and pregnancy outcomes after ovarian stimulation-intrauterine insemination for unexplained infertility. Fertil Steril. 2017 Mar;107(3):756-762.e3. doi: 10.1016/j.fertnstert.2016.12.012. Epub 2017 Jan 12. PMID 28089575
- [Derived] Santoro N, Eisenberg E, Trussell JC, Craig LB, Gracia C, Huang H, Alvero R, Casson P, Christman G, Coutifaris C, Diamond M, Jin S, Legro RS, Robinson RD, Schlaff WD, Zhang H; Reproductive Medicine Network Investigators. Fertility-related quality of life from two RCT cohorts with infertility: unexplained infertility and polycystic ovary syndrome. Hum Reprod. 2016 Oct;31(10):2268-79. doi: 10.1093/humrep/dew175. Epub 2016 Jul 7. PMID 27402910
- [Derived] Hansen KR, He AL, Styer AK, Wild RA, Butts S, Engmann L, Diamond MP, Legro RS, Coutifaris C, Alvero R, Robinson RD, Casson P, Christman GM, Huang H, Santoro N, Eisenberg E, Zhang H; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Predictors of pregnancy and live-birth in couples with unexplained infertility after ovarian stimulation-intrauterine insemination. Fertil Steril. 2016 Jun;105(6):1575-1583.e2. doi: 10.1016/j.fertnstert.2016.02.020. Epub 2016 Mar 3. PMID 26949110
- [Derived] Steiner AZ, Diamond MP, Legro RS, Schlaff WD, Barnhart KT, Casson PR, Christman GM, Alvero R, Hansen KR, Geisler WM, Thomas T, Santoro N, Zhang H, Eisenberg E; Reproductive Medicine Network. Chlamydia trachomatis immunoglobulin G3 seropositivity is a predictor of reproductive outcomes in infertile women with patent fallopian tubes. Fertil Steril. 2015 Dec;104(6):1522-6. doi: 10.1016/j.fertnstert.2015.08.022. Epub 2015 Sep 25. PMID 26413816
- [Derived] Diamond MP, Legro RS, Coutifaris C, Alvero R, Robinson RD, Casson P, Christman GM, Ager J, Huang H, Hansen KR, Baker V, Usadi R, Seungdamrong A, Bates GW, Rosen RM, Haisenleder D, Krawetz SA, Barnhart K, Trussell JC, Ohl D, Jin Y, Santoro N, Eisenberg E, Zhang H; NICHD Reproductive Medicine Network. Letrozole, Gonadotropin, or Clomiphene for Unexplained Infertility. N Engl J Med. 2015 Sep 24;373(13):1230-40. doi: 10.1056/NEJMoa1414827. PMID 26398071
- [Derived] Kuang H, Jin S, Thomas T, Engmann L, Hansen KR, Coutifaris C, Casson P, Christman G, Alvero R, Santoro N, Eisenberg E, Diamond MP, Legro RS, Zhang H; Reproductive Medicine Network. Predictors of participant retention in infertility treatment trials. Fertil Steril. 2015 Nov;104(5):1236-43.e1-2. doi: 10.1016/j.fertnstert.2015.08.001. Epub 2015 Sep 3. PMID 26354094
- [Derived] Diamond MP, Legro RS, Coutifaris C, Alvero R, Robinson RD, Casson P, Christman GM, Ager J, Huang H, Hansen KR, Baker V, Usadi R, Seungdamrong A, Bates GW, Rosen RM, Haisonleder D, Krawetz SA, Barnhart K, Trussell JC, Jin Y, Santoro N, Eisenberg E, Zhang H; National Institute of Child Health and Human Development (NICHD) Reproductive Medicine Network. Assessment of multiple intrauterine gestations from ovarian stimulation (AMIGOS) trial: baseline characteristics. Fertil Steril. 2015 Apr;103(4):962-973.e4. doi: 10.1016/j.fertnstert.2014.12.130. Epub 2015 Feb 20. PMID 25707331
- See also: Reproductive Medicine Network Homepage — http://c2s2.yale.edu/rmn/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH)
Started | 299 | 300 | 301
Completed | 246 | 251 | 249
Not Completed | 53 | 49 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH) | Total
Number analyzed (Participants) | 299 | 300 | 301 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (4.3) | 32.0 (4.6) | 32.2 (4.1) | 32.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 300 | 301 | 900
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 299 | 300 | 301 | 900

OUTCOME MEASURES:

1. Primary Outcome: Multiple Gestation Rate Following Recruitment of Multiple Follicular Development With an AI, as Compared to CC and FSH.
Time Frame: Participants were followed for the duration of their treatment and, if pregnant through 6 weeks post-delivery, up to 66 weeks
Measure: Number; unit: number of multiples
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH)
Number analyzed (Participants) | 85 | 106 | 140
number of multiples | 9 | 8 | 34

2. Secondary Outcome: Rate of Pregnancy Obtained
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH)
Number analyzed (Participants) | 299 | 300 | 301
participants | 85 | 106 | 140

3. Secondary Outcome: Time to Pregnancy
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH)
Number analyzed (Participants) | 299 | 300 | 301
days | 67.2 (55.6) | 67.4 (49.8) | 62.3 (43.8)

4. Secondary Outcome: Live Birth Rate
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH)
Number analyzed (Participants) | 299 | 300 | 301
participants | 56 | 70 | 97

ADVERSE EVENTS:
Description: The Numbers of Participants at Risk are different from the numbers provided in the Participant Flow module as not all subjects who were analyzed were administered study drug and therefore not all subjects were at risk for Adverse Events. Intent-to-treat analysis kept them in the study, but they had no AE risk.
Arm/Group | Aromatase Inhibitors (AI) | Clomiphene Citrate (CC) | Follicle Stimulating Hormone (FSH)
Serious Adverse Events (participants affected / at risk) | 11/291 | 12/298 | 25/297
Other Adverse Events (participants affected / at risk) | 218/291 | 214/298 | 217/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aromatase Inhibitors (AI) (N=291) | Clomiphene Citrate (CC) (N=298) | Follicle Stimulating Hormone (FSH) (N=297)
Presumed Pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pyosalpinx Post IUI (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pain due to ovarian enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy of Unknown Location (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 1 (1)
Acute viral illness (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hemorrhagic Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hospitalization for pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Severe pre-eclampsia; HELLP syndrome, preterm labor (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Emergency C-section due to eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Hospitalization due to shorness of breath; pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Congenital anomaly (Congenital, familial and genetic disorders) | 2 (2) | 3 (3) | 3 (3)
Neonatal Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 5 (5) | 11 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aromatase Inhibitors (AI) (N=291) | Clomiphene Citrate (CC) (N=298) | Follicle Stimulating Hormone (FSH) (N=297)
Abdominal Bloating (Gastrointestinal disorders) | 54 (54) | 50 (50) | 81 (81)
Breast Pain (Reproductive system and breast disorders) | 26 (26) | 19 (19) | 65 (65)
Constipation (Gastrointestinal disorders) | 8 (8) | 28 (28) | 6 (6)
Headache (Nervous system disorders) | 122 (122) | 104 (104) | 89 (89)
Hot Flashes (Endocrine disorders) | 49 (49) | 92 (92) | 25 (25)
Injection Site Reaction (General disorders) | 9 (9) | 6 (6) | 32 (32)
Joint/Limb pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No